CLINICAL TRIAL: NCT02135887
Title: The Purpose of This Study is to Evaluate the Effectiveness of MB-6 as Adjuvant Therapy in Reducing Neutropenia When Given Oxaliplatin-based Chemotherapy in Patients With Stage 3 Colorectal Cancer Previously Treated With Surgery.
Brief Title: A Trial of MB-6 for Reduction of Neutropenia Induced by Chemotherapy in Patients With Stage III Colorectal Cancer.
Acronym: MB-6
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MB104CLCT02
Record Dates: First submitted 2014-05-06; First posted 2014-05-12 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Stage III Colorectal Cancer; Neutropenia
Keywords: Stage III Colorectal Cancer; Grade 4 Neutropenia; MB-6
MeSH Terms: conditions — Colorectal Neoplasms; Neutropenia | interventions — Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MB-6+FOLFOX chemotherapy: MB-6, 6 capsules tid be taken with meals plus FOLFOX chemotherapy, will be given for 18 weeks
  Interventions: Drug: MB-6
- Placebo+FOLFOX chemotherapy: Placebo, 6 capsules tid be taken with meals plus FOLFOX chemotherapy, will be given for 18 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MB-6 — 6# TID with meal
  Other Names: Folinic acid; Fluorouracil ; Oxaliplatin
  Groups: MB-6+FOLFOX chemotherapy
Drug: Placebo — 6# TID with meal
  Other Names: Folinic acid; Fluorouracil ; Oxaliplatin
  Groups: Placebo+FOLFOX chemotherapy

SUMMARY:
This is a randomized, double-blind, placebo-controlled multi-center phaseⅢstudy to evaluate efficacy and safety of oxaliplatin-based chemotherapy plus MB-6(320 mg/capsule, 6 capsules tid) in patients with stage 3 colorectal cancer who underwent surgical excision of their primary tumor.

DETAILED DESCRIPTION:
The investigational new drug, MB-6, in the proposed clinical trial is to be used as an adjuvant therapy for metastatic colorectal cancer patients. All of six extracts have been used in human with a long history, and many literatures reported the medicinal use either individually or as ingredients of formulations. MB-6 may provide its therapeutic benefits via inhibition of tumor induction or enhancing the efficacy of chemotherapy in colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 20 years of age or older.
2. Histologically or cytologically confirmed stage 3 colorectal adenocarcinoma.
3. Complete resection of the primary tumor without gross or microscopic evidence of residual disease.
4. No more than 8 weeks have elapsed from the time of surgery and have recovered from the effects.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) < 2 at the time of screening.
6. Hematological function: ANC≥1500/mm3, Hemoglobin ≥9.0 g/dL, Platelet count ≥100000/mm3.
7. Kidney function:Serum creatinine <2 mg/dL.
8. Liver function: AST ≤3 times ULN, ALT ≤3 times ULN, Total Bilirubin ≤2 times ULN.
9. Ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.
10. Men and women of childbearing potential must agree to employ adequate contraception during the study period.

Exclusion Criteria:

1. History of second primary malignancies except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix.
2. Systemic chemotherapy, immune therapy or experimental or approved antibodies/proteins (e.g. bevacizumab) administered after surgery and prior to randomization.
3. Concurrent treatment with any other anticancer therapy.
4. Radiotherapy ≤14 days prior to randomization.
5. Any unresolved toxicity > CTC (Common Toxicity Criteria) grade 1 from previous anti-cancer therapy (including radiotherapy) except haematological toxicity and alopecia.
6. Patients with congestive heart failure, epilepsy, or other significant medical conditions as judged by the investigator.
7. Contraindications to FOLFOX chemotherapy: peripheral neuropathy NCI CTC >1, liver failure, uncontrolled coronary heart disease, myocardial infarction within the previous 6 months before randomization.
8. Patient of child-bearing potential is evidently pregnant or is breast feeding.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 184 patients with stage III colorectal cancer underwent surgery will be recruited into the study for receiving adjuvant therapy over 18 weeks.
Sampling Method: Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2013-11-04 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the incidence of grade 4 neutropenia during the chemotherapy period, defined as an absolute neutrophil count (ANC) <500/mm3. | 18 weeks
  The primary endpoint is the incidence of grade 4 neutropenia during the chemotherapy, defined as an absolute neutrophil count (ANC)<500/mm3

SECONDARY OUTCOMES:
Time to first Grade 4 Neutropenia | 18 weeks
  To determine the time interval from randomization to the first episode of grade 4 Neutropenia.
  The analyses for incidence of study event will be conducted using logistic regression model method to adjust for gender and the regimen of chemotherapy (e.g., FOLFOX4 or FOLFOX6).
Incidence of Febrile Neutropenia | 18 weeks
  The febrile neutropenia is defined as an ANC <1000/mm3 and a single temperature ≥38.3 degree of C or a sustained temperature of ≥38.0 degree C for more than one hour.
Incidence of Grade 3 or 4 Neutropenia | 18 weeks
  The grade 3 or 4 neutropenia during the chemotherapy period is defined as an absolute neutrophil count (ANC) <1000/mm3.
Change in Serum Creatinine level | 18 weeks
  Any change in Serum Creatinine level during the chemotherapy period
Health-Related Quality of Life (HRQoL) - QLQ-C30 | 18 weeks
  Health-Related Quality of Life (HRQoL) - QLQ-C30 should be completed at baseline, day 71 and end of study.
Quality of Life -VAS on Fatigue, Constipation, Appetite | 18 weeks
  Quality of Life -VAS on Fatigue, Constipation, Appetite will be assessed by patients every two weeks until end of study.
Compliance with Chemotherapy | 18 weeks
  The compliance with chemotherapy will be summarized by descriptive statistic and listed by each cycle and overall period.
Increase in Body Weight | 18 weeks
  Any increased body weight during the chemotherapy period.

CONTACTS AND LOCATIONS:
Overall Officials: William Chen, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- Microbio Co., Ltd., Taipei, Taiwan